CLINICAL TRIAL: NCT05144919
Title: The Role of Agricultural Biodiversity in Thet Diet: a Vietnamese Study
Brief Title: Biodiversity in the Diet in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: HealthBridge (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015/1205
Record Dates: First submitted 2021-12-02; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Biodiversity; Food Intake; Nutritional Status
Keywords: Biodiversity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The control group will continue to receive routine health check and nutrition education from health staff at commune health facilities. Access to agriculture extension services as offered by provincial staff will also continue as normal.
- Intervention (Experimental): The intervention group will receive capacity building sessions on both Agriculture and Nutrition, in addition to access to routine health and nutrition checks, and agriculture extension as offered by commune and provincial staff as normal.
  Interventions: Behavioral: Promotion of a biodiverse diet

INTERVENTIONS:
Behavioral: Promotion of a biodiverse diet — Component 1 - Participatory Identification of Intervention Approach (PIIA) Component 2. Local stakeholder consultation Component 3. Sensitisation of community Diversity club will receive capacity building from a Village health worker based on the prioritised species selected in component 2.
  The following topics will be covered for each species selected for promotion:
  1. Where to locally source inputs and expected price
  2. How/when to prepare plots using organic inputs
  3. Planting and best-practice management practices
  4. Seed saving and storage
  5. Possible intercropping combinations OR ecosystem services provided Component 4. Active Cooking demonstrations and Nutrition Education and counselling: Diversified cooking practices
  Arms: Intervention

SUMMARY:
Agricultural biodiversity can have an important role in improving diet diversity, quality and nutrition and can be seen as the foundation of the food and nutrition value chain. Increasing the availability and access to local agricultural and/or wild biodiversity genetic resources has the potential to increase production, making more food available for consumption as long as entitlements to access it exist. However, as the history of food security interventions has shown, increasing the production and supply of staple crops alone is not enough to improve food security or nutritional status. However, while agricultural diversification is an important component, it is not alone sufficient to improve diet diversity. Other system elements including women's education and knowledge, intra-household dynamics and women's status and cultural beliefs and practices that improves children's health and nutrition are important to ensure biodiversity has a successful role in improving dietary diversity and quality.

ELIGIBILITY:
Inclusion Criteria:

* villages: Characterized as Thai village. Only Thai villages will be selected for the study as agriculture practices, diets, food preferences, language and cultures can change drastically between ethnic groups.
* participants: i) Woman of reproductive age (between 15-49 years) who are the mother or primary caregiver of a child between 12 and 23 months of age. This age group is part of the critical 1000 day window for child development and marks the time when young children can potentially consume all foods from the household pot and consume a more diverse diet. As such, it is from this age group that biodiversity can have an effect on children's diets.

ii) Both the woman and the child should be permanent residents in the village selected and do not temporarily migrate outside the village cluster during the year.

Exclusion Criteria:

* villages: Urban center of commune/province as these villages/cities do not have agriculture or home garden opportunities
* participants: currently engaged in other agriculture or nutrition programme or intervention apart from what is offered by government extension workers

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Consumption of nutrient rich food groups | 24 months
  Mean intakes (g) of Dark Green leafy vegetables, Vitamin A Rich Fruit and Vegetable and Legumes, nuts and seeds by mothers and young children.
Consumption of nutrient rich food groups | 24 months
  Proportion of women and children consuming 3 Dark Green leafy vegetables, Vitamin A Rich Fruit and Vegetable and Legumes, nuts and seeds by mothers and young children.
dietary quality | 24 months
  Proportion of women and children reaching estimated average requirement (EAR) of iron and vitamin A
Mean species richness consumed | 24 months
  Mean species richness consumed

SECONDARY OUTCOMES:
Food and nutrient intake | 24 months
  Proportion of women and children reaching EAR of 16 key nutrients
Nutritional Knowledge of Women | 24 months
  Mean score from a set of nutrient and food specific questions
Individual Dietary Diversity Score | 24 months
  Individual Dietary Diversity Score by women and children
Minimum Dietary Diversity | 24 months
  Proportion of women and children that consumed 5 or more food groups (out of 10)
nutritional status | 24 months
  Mean change from baseline in height-for-age Z-scores Mean change from baseline in weight-for-height Z-scores
Women's Empowerment | 24 months
  Decision making power on selection of species to cultivate, use at homestead and time spent
Consumption of processed foods and drinks | 24 months
  Mean daily intakes (g) of processed foods and drinks Mean proportion of daily energy, fat, salt and sugar intakes from processed foods
income | 24 months
  Household Income from sale of home garden species, agriculture, off-farm employment

CONTACTS AND LOCATIONS:
Locations (1):
- Mai Sơn, Sơn La Province, Vietnam

REFERENCES:
- See also: Related Info — http://www.bioversityinternational.org/